CLINICAL TRIAL: NCT04885712
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of Pioglitazone 15mg or Pioglitazone 30mg Add-on in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin and Dapagliflozin
Brief Title: A Study to Evaluate the Efficacy and Safety of Pioglitazone 15mg or 30mg Add-on in Patients With Type 2 Diabetes Mellitus Inadequately Controlled With Metformin and Dapagliflozin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR-DPC-CT-301
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Pioglitazone; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Metformin≥1000mg + Dapagliflozin 10mg + Pioglitazone 15mg + Pioglitazone 30mg Placebo (Experimental): Metformin≥1000mg Dapagliflozin 10mg Pioglitazone 15mg Pioglitazone 30mg placebo
  Interventions: Drug: Metformin≥1000mg; Drug: Pioglitazone 15mg; Drug: Pioglitazone 30mg Placebo; Drug: Dapagliflozin 10mg
- Metformin≥1000mg + Dapagliflozin 10mg + Pioglitazone 30mg +Pioglitazone 15mg Placebo (Experimental): Metformin≥1000mg Dapagliflozin 10mg Pioglitazone 30mg Pioglitazone 15mg placebo
  Interventions: Drug: Metformin≥1000mg; Drug: Pioglitazone 30 mg; Drug: Pioglitazone 15mg Placebo; Drug: Dapagliflozin 10mg
- Metformin≥1000mg + Dapagliflozin 10mg + Pioglitazone 15mg Placebo+ Pioglitazone 30mg Placebo (Active Comparator): Metformin≥1000mg Dapagliflozin 10mg Pioglitazone 15mg placebo Pioglitazone 30mg placebo
  Interventions: Drug: Metformin≥1000mg; Drug: Pioglitazone 15mg Placebo; Drug: Pioglitazone 30mg Placebo; Drug: Dapagliflozin 10mg

INTERVENTIONS:
Drug: Metformin≥1000mg — Subjects take the investigational products once a day for 24 weeks.
  Other Names: BR3003D
Drug: Pioglitazone 15mg — Subjects take the investigational products once a day for 24 weeks.
  Other Names: BR3003A-1
  Arms: Metformin≥1000mg + Dapagliflozin 10mg + Pioglitazone 15mg + Pioglitazone 30mg Placebo
Drug: Pioglitazone 30 mg — Subjects take the investigational products once a day for 24 weeks.
  Other Names: BR3003B-1
  Arms: Metformin≥1000mg + Dapagliflozin 10mg + Pioglitazone 30mg +Pioglitazone 15mg Placebo
Drug: Pioglitazone 15mg Placebo — Subjects take the investigational products once a day for 24 weeks.
  Other Names: BR3003A-2
  Arms: Metformin≥1000mg + Dapagliflozin 10mg + Pioglitazone 15mg Placebo+ Pioglitazone 30mg Placebo; Metformin≥1000mg + Dapagliflozin 10mg + Pioglitazone 30mg +Pioglitazone 15mg Placebo
Drug: Pioglitazone 30mg Placebo — Subjects take the investigational products once a day for 24 weeks.
  Other Names: BR3003B-2
  Arms: Metformin≥1000mg + Dapagliflozin 10mg + Pioglitazone 15mg + Pioglitazone 30mg Placebo; Metformin≥1000mg + Dapagliflozin 10mg + Pioglitazone 15mg Placebo+ Pioglitazone 30mg Placebo
Drug: Dapagliflozin 10mg — Subjects take the investigational products once a day for 24 weeks.
  Other Names: BR3003C

SUMMARY:
A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of Pioglitazone 15mg or Pioglitazone 30mg Add-on in Patients with Type 2 Diabetes Mellitus Inadequately Controlled with Metformin and Dapagliflozin

ELIGIBILITY:
Inclusion Criteria:

1. Those who voluntarily signed the informed consent to participate in this study.
2. Adults aged 19 years or older.
3. Those diagnosed with type 2 diabetes mellitus.
4. Subjects taking constant doses of ≥1000mg of Metformin and 10 mg of Dapagliflozin for more than 8 weeks at Visit 1 (regardless of dosage forms (immediate-release and sustained-release) and single agent or combination drug.)
5. Subjects with 7% ≤ HbA1c ≤ 10.5% at Visit 1 and Visit 2
6. Subjects able to understand the study, comply with study procedures, and attend all scheduled visits.

Exclusion Criteria:

1. Uncontrolled hyperglycemia at Visit 1 or Visit 2 (subjects with FPG > 270 mg/dL as a result of the test conducted by the study institution.)
2. Medication compliance is <70% or >120% for each BR3003D, BR3003C, BR3003A-2, and BR3003B-2 during the Run-in period at Visit 2.
3. Patients with other types of diabetes instead of type 2 diabetes (e.g., type 1 diabetes, secondary diabetes, or congenital renal glycosuria).
4. Patients with uncontrolled, severe diabetic complications (e.g., proliferative diabetic retinopathy uncontrolled despite medication and severe diabetic neuropathy)
5. Those who suffered from acute or chronic metabolic acidosis within 3 months as of Visit 1, including lactic acidosis and diabetic ketoacidosis.
6. Those with > 40 kg/m2 of BMI measured at Visit 1.
7. Those with uncontrolled hypertension at Visit 1 or Visit 2 (SBP > 180 mmHg or DBP > 110 mmHg).
8. Those diagnosed with cardiovascular diseases (myocardial infarction, stroke, unstable angina, and transient ischemic attack (TIA)) or undergo revascularization within 3 months as of Visit 1
9. Those with heart failure (NYHA class II~IV) or who had suffered from heart failure.
10. Those who suffered from gastrointestinal diseases that may affect the absorption, distribution, metabolism, and excretion of investigational products or had underwent surgery;
11. Those who underwent surgery requiring general anesthesia within 4 weeks as of Visit 1 or who are scheduled to receive such surgery within 4 weeks after the study ends
12. Those with a history of malignant tumor within 5 years as of Visit 1
13. Those who have a clinically significant liver disease
14. Those who have a clinically significant renal disease
15. Those with clinically significant hematuria detected at Visit 1 or Visit 2
16. Those with chronic diseases requiring the continued use of systemic steroid or immunosuppressants (oral administration, injection, or inhalation).
17. Patients with pituitary insufficiency or adrenal insufficiency.
18. Those with clinically significant severe infection or trauma based on an investigator's judgement.
19. Patients with AIDS.
20. Patients with acute or chronic diseases that may cause histotoxic hypoxia such as respiratory failure and shock.
21. Those who need treatment due to dehydration caused by persistent diarrhea and vomiting or at a risk of fluid volume depletion.
22. Those who have been administered with the following drugs or expected to require the continued administration during the study period:

    * Those administered with systemic steroid agents (Prednisolone, >30 mg/day) within 2 weeks as of Visit 1.
    * Those being administered with thyroid medications and whose dose has been modified within 6 weeks as of Visit 1 (however, dose reduction is accepted.)
    * Those being administered with diuretics and whose dose has been modified within 8 weeks as of Visit 1 however, dose reduction is accepted.)
    * Those who have been administered with antidiabetics other than Metformin and Dapagliflozin within 8 weeks as of Visit 1.
    * Those who have been administered with obesity drugs (e.g., phentermine, phendimetrazine, diethylpropion, and mazindol) within 12 weeks as of Visit 1.
    * Those who need to take prohibited concomitant medications stated here during the study period.
23. Those with history of alcohol or drug abuse within 1 year as of Visit 1.
24. Those who had allergic reaction to main ingredients or components of the investigational products.
25. Those who had genetic disorders such as galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption.
26. Females who are pregnant or breastfeeding.
27. Patients planning to become pregnant or of childbearing potential, but not using any recognized contraceptive method
28. Those who are currently participating in other ongoing clinical studies or those who have taken the investigational products from other clinical studies within 12 weeks as of Visit 1
29. Those who are judged unsuitable for the study by a principal investigator or investigators.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c | 24th week
  Changes in HbA1c at the 24th week after the administration of investigational products from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Woo-je Lee, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho YK, Kim KS, Lee BW, Hong JH, Yu JM, Lim S, Kim YA, Lee CB, Kim SS, Kwak SH, Lee WJ. Efficacy and Safety of Pioglitazone Add-on in Patients with Type 2 Diabetes Mellitus Inadequately Controlled with Metformin and Dapagliflozin: A Multicenter, Randomized, Double-blind, and Placebo-controlled Study. Clin Ther. 2024 Sep;46(9):662-669. doi: 10.1016/j.clinthera.2024.06.023. Epub 2024 Jul 26. PMID 39068060